CLINICAL TRIAL: NCT03880565
Title: Advanced REperfusion STrategies for Refractory Cardiac Arrest (The ARREST Trial)
Brief Title: Advanced Reperfusion Strategies for Refractory Cardiac Arrest
Acronym: ARREST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: For early efficacy
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CV-2018-27226
Record Dates: First submitted 2019-03-11; First posted 2019-03-19 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Arrest; Extracorporeal Membrane Oxygenation Complication; Ventricular Fibrillation; Pulseless Ventricular Tachycardia; Out-Of-Hospital Cardiac Arrest
Keywords: advanced reperfusion; mechanical cardiopulmonary resuscitation
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation; Out-of-Hospital Cardiac Arrest | interventions — Extracorporeal Membrane Oxygenation; Resuscitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- ECMO Facilitated Resuscitation (Experimental): Regardless of whether return of spontaneous circulation (ROSC) has been achieved and with on-going mechanical CPR, patients will enter the Cardiac Catheterization Laboratory (CCL) for expeditious VAECMO initiation, if required, followed by coronary angiography and percutaneous coronary intervention (PCI) when appropriate.
  Interventions: Device: Early Extracorporeal Membrane Oxygenation (ECMO) Facilitated Resuscitation
- Standard ACLS Resuscitation (Other): Patients with refractory VF/VT OHCA will be treated with ACLS resuscitation for at least 15 minutes after arrival in the emergency department (ED), or up to 60 minutes from 911 call, after which the physician (MD) can continue resuscitation efforts until ROSC is achieved or futility has been reached based on their clinical judgment. If the patient has not achieved ROSC during the times mentioned above, the ED MD can declare death when he or she believes that ACLS is futile. If ROSC is present upon arrival or has been achieved anytime during resuscitation in the ED, the patient will be taken to the cardiac catheterization laboratory (CCL) for coronary angiography and PCI, and potential VA ECMO or other circulatory support device initiation, as clinically indicated.
  Interventions: Device: Standard Advanced Cardiac Life Support (ACLS) Resuscitation

INTERVENTIONS:
Device: Early Extracorporeal Membrane Oxygenation (ECMO) Facilitated Resuscitation — Early use of ECMO
  Arms: ECMO Facilitated Resuscitation
Device: Standard Advanced Cardiac Life Support (ACLS) Resuscitation — Standard life support resuscitation
  Arms: Standard ACLS Resuscitation

SUMMARY:
This is a Phase II, single center (Under the Center for Resuscitation Medicine at the University of Minnesota Medical School), partially blinded, prospective, intention to treat, safety and efficacy clinical trial, randomizing adult patients (18-75 years old) with refractory ventricular fibrillation/pulseless ventricular tachycardia (VF/VT) out-of hospital cardiac arrest (OHCA) who are transferred by emergency medical services (EMS) with ongoing mechanical cardiopulmonary resuscitation (CPR) or who are resuscitated to receive one of the 2 local standards of care practiced in our community: 1) Early Extracorporeal Membrane Oxygenation (ECMO) Facilitated Resuscitation or 2) Standard Advanced Cardiac Life Support (ACLS) Resuscitation

ELIGIBILITY:
Inclusion Criteria:

* Adults (presumed or known to be aged 18-75 years, inclusive),
* An initial documented OHCA rhythm of VF/VT,
* No ROSC following 3 defibrillation shocks,
* Body morphology able to accommodate a Lund University Cardiac Arrest System (LUCAS™) automated CPR device, and
* Estimated transfer time from the scene to the ED or CCL of < 30 minutes.

Exclusion Criteria:

* Age < 18 years old or > 75 years old;
* Non-shockable initial OHCA rhythm (pulseless electrical activity [PEA] or asystole);
* Valid do-not-attempt-resuscitation orders (DNAR);
* Blunt, penetrating, or burn-related injury, drowning, electrocution or known overdose;
* Known prisoners;
* Known pregnancy;
* Nursing home residents;
* Unavailability of the cardiac catheterization laboratory.
* Severe concomitant illness that drastically shortens life expectancy or increases risk of the procedure;
* Absolute contraindications to emergent coronary angiography including known anaphylactic reaction to angiographic contrast media and/or active gastrointestinal or internal bleeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2020-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Demetris Yannopoulos, MD, Principal Investigator — University of Minnesota; Tom Aufderheide, MD, Study Chair — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yannopoulos D, Bartos J, Raveendran G, Walser E, Connett J, Murray TA, Collins G, Zhang L, Kalra R, Kosmopoulos M, John R, Shaffer A, Frascone RJ, Wesley K, Conterato M, Biros M, Tolar J, Aufderheide TP. Advanced reperfusion strategies for patients with out-of-hospital cardiac arrest and refractory ventricular fibrillation (ARREST): a phase 2, single centre, open-label, randomised controlled trial. Lancet. 2020 Dec 5;396(10265):1807-1816. doi: 10.1016/S0140-6736(20)32338-2. Epub 2020 Nov 13. PMID 33197396

RESULTS

PARTICIPANT FLOW:
Groups:
- ECMO Facilitated Resuscitation: Early Extracorporeal Membrane Oxygenation (ECMO) Facilitated Resuscitation: ECMO is initiated expeditiously, regardless of whether return of spontaneous circulation (ROSC) has been achieved and with on-going mechanical CPR, if required, followed by coronary angiography and percutaneous coronary intervention (PCI) when appropriate.
  Early Extracorporeal Membrane Oxygenation (ECMO) Facilitated Resuscitation: Early use of ECMO
- Standard ACLS Resuscitation: Standard Advanced Cardiac Life Support (ACLS) Resuscitation: Patients with refractory VF/VT OHCA will be treated with ACLS resuscitation for at least 15 minutes after arrival in the emergency department (ED), or up to 60 minutes from 911 call, after which the physician (MD) can continue resuscitation efforts until ROSC is achieved or futility has been reached based on their clinical judgment. If the patient has not achieved ROSC during the times mentioned above, the ED MD can declare death when he or she believes that ACLS is futile. If ROSC is present upon arrival or has been achieved anytime during resuscitation in the ED, the patient will be taken to the cardiac catheterization laboratory (CCL) for coronary angiography and PCI and potential VA ECMO or other circulatory support device initiation, as clinically indicated.
  Standard Advanced Cardiac Life Support (ACLS) Resuscitation: Standard life support resuscitation
Period: Overall Study
Arm/Group | ECMO Facilitated Resuscitation | Standard ACLS Resuscitation
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ECMO Facilitated Resuscitation | Standard ACLS Resuscitation | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (9.7) | 57.1 (10.6) | 58.5 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 14 | 11 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 6 | 2 | 8
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 12 | 18
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Survival
Description: Number of participants who survived to hospital discharge
Time Frame: Approximately 25 days
Measure: Count of Participants; unit: Participants
Arm/Group | ECMO Facilitated Resuscitation | Standard ACLS Resuscitation
Number analyzed (Participants) | 15 | 15
Participants | 6 | 1

2. Secondary Outcome: Modified Rankin Scale (mRS) Score
Description: mRS scale ranges from 0 (no residual symptoms) to 6 (dead). Scores of 3 (the patient has moderate disability), 2 (the patient has slight disability), 1 (the patient has no significant disability), and 0 indicate favorable outcome. Higher scores on the scale indicate more severe disability. Outcome is reported as the mean score. Outcome is collected and reported at hospital discharge (average of 25 days) and at three and six months following.
Time Frame: At hospital discharge (average of 25 days), 3 months, 6 months
Population: All participants who completed each time point are included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ECMO Facilitated Resuscitation | Standard ACLS Resuscitation
Number analyzed (Participants) | 15 | 15
score on a scale
  Hospital Discharge: number analyzed (Participants) | 6 | 1
  Hospital Discharge | 3.8 [3 to 4.6] | 5 [NA to NA] — There is only one participant in this group.
  Three Months: number analyzed (Participants) | 6 | 0
  Three Months | 2 [.9 to 3.4] |
  Six Months: number analyzed (Participants) | 6 | 0
  Six Months | 1.5 [.4 to 2.6] |

3. Secondary Outcome: Cerebral Performance Categories (CPC) Scale
Description: CPC scale ranges from 1 (good cerebral performance) to 5 (brain death). CPC scores of 2 (moderate cerebral disability) and 1 indicate functional status. Higher scores on the scale indicate worse cerebral performance. Outcome is reported as the mean score. Outcome is collected and reported at hospital discharge (average of 25 days) and at three and six months following.
Time Frame: At hospital discharge (average of 25 days), 3 months, 6 months
Population: All participants who completed each time point are included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | ECMO Facilitated Resuscitation | Standard ACLS Resuscitation
Number analyzed (Participants) | 15 | 15
score on a scale
  Hospital Discharge: number analyzed (Participants) | 6 | 1
  Hospital Discharge | 2.5 [1.9 to 3.1] | 4 [NA to NA] — There is only one participant in this group.
  Three Months: number analyzed (Participants) | 6 | 0
  Three Months | 1.2 [.7 to 1.6] |
  Six Months: number analyzed (Participants) | 6 | 0
  Six Months | 1.2 [.7 to 1.6] |

4. Secondary Outcome: Treatment Cost
Description: Outcome is reported as the mean treatment cost in dollars.
Time Frame: 6 months
Population: Outcome was not collected.
Arm/Group | ECMO Facilitated Resuscitation | Standard ACLS Resuscitation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Six months following hospital discharge
Arm/Group | ECMO Facilitated Resuscitation | Standard ACLS Resuscitation
All-Cause Mortality (participants affected / at risk) | 9/15 | 14/15
Serious Adverse Events (participants affected / at risk) | 15/15 | 15/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECMO Facilitated Resuscitation (N=15) | Standard ACLS Resuscitation (N=15)
Bleeding (Blood and lymphatic system disorders) | 7 (7) | 0 (0)
Circulatory Disorder (Blood and lymphatic system disorders) | 15 (45) | 15 (20)
Central Nervous System Disorders (Nervous system disorders) | 9 (12) | 1 (3)
CPR Trauma (Injury, poisoning and procedural complications) | 11 (198) | 1 (2)
Endocrine Disorders (Endocrine disorders) | 13 (20) | 10 (12)
Gastrointestinal Disorder (Gastrointestinal disorders) | 9 (10) | 2 (2)
Infection (Infections and infestations) | 5 (6) | 0 (0)
Kidney Disorders (Renal and urinary disorders) | 10 (18) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 2 (4)
Other Disorder (General disorders) | 9 (13) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03880565/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT03880565/ICF_000.pdf